CLINICAL TRIAL: NCT00052637
Title: An Open, Comparative, Within Patient, Controlled Phase III, Multicenter Study Of HEXVIX Fluorescence Cystoscopy And White Light Cystoscopy In the Detection Of Carcinoma In Situ In Patients With Bladder Cancer
Brief Title: Cystoscopy and Hexyl 5-Aminolevulinate in Detecting Carcinoma In Situ in Patients With Bladder Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Photocure (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Diagnostic
Other Study IDs: PC B301/01; UCLA-0201058; CDR0000258579 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-10

CONDITIONS: Bladder Cancer
Keywords: bladder cancer; recurrent bladder cancer; stage 0 bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — 5-aminolevulinic acid hexyl ester; Biopsy; Cystoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: hexaminolevulinate
Procedure: biopsy
Procedure: cystoscopy

SUMMARY:
RATIONALE: Diagnostic procedures such as cystoscopy may improve the ability to detect cancer and to determine the extent of disease.

PURPOSE: Diagnostic trial to compare the effectiveness of cystoscopy using hexyl 5-aminolevulinate and two light sources in detecting carcinoma in situ in patients who have bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare blue light fluorescent cystoscopy with reconstituted hexyl 5-aminolevulinate (Hexvix®) vs white light cystoscopy for the detection of carcinoma in situ (CIS) in patients with bladder cancer.
* Compare the positive and false detection rates of histologically confirmed non-CIS lesions and dysplasia by these modalities in these patients.
* Compare the false detection rate of histologically confirmed CIS lesions by these modalities in these patients.
* Compare the number of tumor lesions and dysplasia detected by these modalities in these patients.
* Compare management of patients after evaluation with these modalities.
* Determine the safety of reconstituted hexyl 5-aminolevulinate (Hexvix®) in these patients.

OUTLINE: This is an open-label, multicenter study.

Patients undergo bladder catheterization and instillation of reconstituted hexyl 5-aminolevulinate (Hexvix®). After 60 minutes the bladder is evacuated, and the patient undergoes cystoscopic examination of the bladder by white light and then blue light fluorescence. Biopsies are taken of all suspicious areas seen under white and/or blue light modalities, and one normal-appearing area seen under both light modalities, and papillary lesions are resected.

Patients are followed at 7 days after procedure.

PROJECTED ACCRUAL: A total of 420 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Indication for cystoscopy for suspected or confirmed bladder cancer
* Meets at least one of the following criteria:

  * Multiple bladder lesions
  * Bladder lesion greater than 3 cm
  * Bladder tumor of at least stage T1
  * Grade 2 or 3 bladder tumor
  * Recurrent bladder cancer
* No positive cytology obtained in the last 4 weeks
* No prior G3 tumor with one set of positive random biopsies
* No porphyria

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* No gross hematuria

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 1 month after study
* No known allergy to reconstituted hexyl 5-aminolevulinate or a similar compound
* No concurrent condition that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 3 months since prior BCG

Chemotherapy

* More than 3 months since prior chemotherapy

  * Single prior dose of chemotherapy for prevention of seeding after resection allowed

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* More than 30 days since prior participation in another clinical trial
* No concurrent participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-09; Primary Completion 2002-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schulam, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States